CLINICAL TRIAL: NCT03283332
Title: Determinants of Adolescent Social Well-being and Health: a London Based Longitudinal Study of Young People From Different Ethnic Groups
Brief Title: Determinants of Adolescent, Now Young Adults, Social Well-being and Health: Longitudinal Follow-up
Acronym: DASH
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Medical Research Council (Other Government); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Other Study IDs: 05/MRE10/43
Record Dates: First submitted 2017-09-08; First posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Cardiovascular Risk Factor
Keywords: Ethnicity; adolescents; cohort; longitudinal; health inequalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
Black and ethnic minority groups living in the UK experience high rates of chronic diseases such as diabetes, hypertension and heart disease, general morbidity and poor mental health. The cause of these excess rates is unknown but obesity, smoking, diet and deprivation are important contributing factors. There is also global evidence of the association of these diseases in adulthood with health and deprivation in early life and childhood. Persisting social deprivation over the lifecourse is disproportionately borne by some ethnic minorities (Harding and Balarajan 2001) but the impact on the health of their children is virtually unknown. Least is known about the health of Black Caribbean young people. It is important to examine risk factor differences by social predictors within the ethnic minority groups as well as between them. The DASH Study started as a school-based cohort study of adolescents from the main ethnic groups (White British, Black Caribbean, Black African, Indian, Pakistani and Bangladeshi) in 10 London boroughs. Wave 1 took place in 2002/03 (MREC Ref: MREC/2/10/12), when participants were aged 11-13 years (school years 7 and 8). Wave 2 took place in 2005/06 (MREC Ref: 05/MRE10/43) when they were 14-16 years (school years 9 and 10). Wave 3 took place in 2010/2011, when participants were aged 19-21 years and involved a postal follow-up complemented by telephone interview and on-line questionnaires. The current proposal is for a feasibility study, using a small sample of the DASH cohort, to inform the design of the next full face-to-face follow-up. DASH will be the first large scale UK longitudinal cohort of ethnic minority youths with both social and biological measures from childhood to early adulthood. It will allow detailed examination of ethnic differences in the social patterning of biological mechanisms and pre-clinical disease in young adulthood.

DETAILED DESCRIPTION:
Background:

Black and ethnic minority groups living in the UK experience high rates of chronic diseases such as diabetes, hypertension and heart disease, general morbidity and poor mental health. The cause of these excess rates is unknown but obesity, smoking, diet and deprivation are important contributing factors. There is also global evidence of the association of these diseases in adulthood with health and deprivation in early life and childhood. Persisting social deprivation over the lifecourse is disproportionately borne by some ethnic minorities (Harding and Balarajan 2001) but the impact on the health of their children is virtually unknown. Least is known about the health of Black Caribbean young people. It is important to examine risk factor differences by social predictors within the ethnic minority groups as well as between them. The DASH Study started as a school-based cohort study of adolescents from the main ethnic groups (White British, Black Caribbean, Black African, Indian, Pakistani and Bangladeshi) in 10 London boroughs. Wave 1 took place in 2002/03 (MREC Ref: MREC/2/10/12), when participants were aged 11-13 years (school years 7 and 8). Wave 2 took place in 2005/06 (MREC Ref: 05/MRE10/43) when they were 14-16 years (school years 9 and 10). Wave 3 took place in 2010/2011, when participants were aged 19-21 years and involved a postal follow-up complemented by telephone interview and on-line questionnaires. The current proposal is for a feasibility study, using a small sample of the DASH cohort, to inform the design of the next full face-to-face follow-up. DASH will be the first large scale UK longitudinal cohort of ethnic minority youths with both social and biological measures from childhood to early adulthood. It will allow detailed examination of ethnic differences in the social patterning of biological mechanisms and pre-clinical disease in young adulthood.

Aims:

(i) To conduct a feasibility study to establish the best methods for data collection, including the collection of physical and biological measurements, for subsequent face to face follow-up of the entire cohort.

(ii) To generate a proposal for subsequent follow-up of the entire cohort for submission to MRC, dependent on the findings of the postal and telephone surveys and proposed feasibility study.

Objectives:

I. What are the advantages and disadvantages of conducting the study in the two settings - GP surgeries and homes?

1. Do participants' response rates vary by setting?
2. What are the challenges faced by the nurses in clinics and home visits?
3. Will the quality of data collected (e.g. extent of missing data) vary by setting?
4. Will the delivery of blood samples to the laboratory be reasonably straight forward in each setting? II. What percentage of participants will agree to undertake bio-marker measures? III. Are mental health measures for this age group, typically used with White European populations, culturally appropriate? IV. How will DASH participants' view feedback on their medical results (e.g. blood pressure, weight, blood lipids)? V. Were participants satisfied with the different components of the survey process - contact, consent, data collection? VI. What is the estimated length of time and the resources required for subsequent full follow-up of DASH study members?

Outcome measures:

These will be examined by setting (home visit, GP surgery) using a mixture of quantitative and qualitative methods and are as follows:

I. Percentage response rates - overall, per item/physical measure; II. Percentage consistency of answers to questionnaire items; III. Percentage physical measures within expected range e.g. spirometric measures; IV. Mean length of time for interview; V. Mean length of time for taking physical/biological measures; VI. Qualitative appraisal of cultural appropriateness of mental health measures and of respondents' satisfaction with survey processes.

Sample At the recent telephone survey, respondents were asked if they would be willing to take part in a small feasibility study to prepare for a later full face to face follow-up. Almost all agreed and of those, a sample of 300 (40-50 in each of the main ethnic groups- White British, Black Caribbean, Black African, Pakistani, Bangladeshi, Indian) will be invited to complete a questionnaire, and have physical and physiological measures taken. Interviews will be conducted in respondents' own homes or GP surgeries dependent on the preference of the respondent. As this is a feasibility study, the sample size has been chosen pragmatically to give a reasonable spread, with equal gender representation across the 10 London boroughs that the whole sample was in at wave 2.

Specially trained nurses will conduct the survey in homes or General Practitioners' surgeries, supervised by a nurse manager in the General Practice Research Framework. Nurses will be attached either to the General Research Practice Framework or the Primary Care Research Network.

Main Questionnaire The content reflects mainly questions that were asked in previous waves (general health; health behaviours; psychological well-being; SEC; social support; and relationship with parents). New items include parenthood; age appropriate mental health measures; own education, economic activity and occupation; job strain; caring; 'romantic' relationships; positive and negative emotions; views on their parents being invited to participate in DASH in order to examine generational influences. The investigators will explore two methods of delivery of the questionnaires - self complete questionnaires done prior to visit and computer assisted interviews. If the questionnaire is not completed by the time of the interview, respondents will be asked if they would like to complete a computer assisted interview. Completion of the questionnaire is expected to take about 40 minutes.

Physical/physiological measures As in waves 1/and 2, height, weight, arm, waist and hip circumference, lung function, blood pressure will be measured.

New measures include:

(i)Hand to foot bio-impedance (ii) Bio-markers - HbA1c, total cholesterol, HDL-cholesterol (iii) Dietary assessment - 24 hour recall interviews Qualitative assessment - focus groups and semi-structured interviews. For the new mental health/cognitive measures, the investigators will conduct focus group vignette assessment, based on explanatory model and illness perception theories. This will be carried out in a small sub-sample (6 participants per ethnic group and allowing for 2 gender-specific groups; n=48). Analysis of these data will focus on narratives about the signs and symptoms of different aspects of mental health in the different ethnic groups. These data will provide valuable insights about the appropriateness of measures, usually validated with European populations, for ethnic minority groups.

A research scientist will conduct semi-structured interviews with respondents to obtain feedback on the process of follow-up - what worked well, how best to improve the process, what was un/acceptable etc. The investigators will also enquire about the usefulness of feedback of results. A similar evaluation will take place with the nurses with the aim of identifying best practice in clinics and homes.

Data analysis Descriptive statistics will be used to look at the general distributions and quality of the data collected. Outcomes measured as rates will be examined by data collection setting (GP surgeries vs. home visits), ethnic group and socio-demographic characteristics using standard comparisons technique such as Chi-square test or logistic regression. Mean length of time and any continuous outcomes will be compared using linear regression. In addition, although the sample size of each ethnic group is small, the total sample will allow analyses of the potential social patterning of biological mechanisms in a diverse sample in young adulthood.

ELIGIBILITY:
Inclusion Criteria:

* provision of informed consent

Exclusion Criteria:

* none

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: School children, aged 11-13 years, representing the main UK ethnic groups (White-European, Black African, Black Caribbean, Indian, Pakistani/Bangladeshi, Other, mainly mixed race).
Sampling Method: Probability Sample
Enrollment: 6643 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2012-12-01 (Actual); Study Completion 2012-12-01 (Actual)

PRIMARY OUTCOMES:
Response rate | Through study completion, on average 10 years
  Percentage response rates - overall, per item/physical measure
Interview duration | Through study completion, on average 10 years
  Mean length of time for interview
physical measures duration | Through study completion, on average 10 years
  Mean length of time for physical/biological measures

SECONDARY OUTCOMES:
Weight | Through study completion, on average 10 years
  Body weight, kg
Height | Through study completion, on average 10 years
  Height, cm
waist circumference | Through study completion, on average 10 years
  Waist circumference, cm
blood pressure | Through study completion, on average 10 years
  systolic and diastolic blood pressure, mmHg
Body fat | Through study completion, on average 10 years
  body fat measured by bioelectrical impedence, %
HbA1c | Through study completion, on average 10 years
  Glycated haemoglobin, %
Total cholesterol | Through study completion, on average 10 years
  Serum total cholesterol, mmol/l
HDL-cholesterol | Through study completion, on average 10 years
  Serum high-density-lipoprotein cholesterol, mmol/l
Energy intake | Through study completion, on average 10 years
  Dietary energy intake, kcal/day
Fat intake | Through study completion, on average 10 years
  Dietary fat intake, % of total energy intake
Saturated fat intake | Through study completion, on average 10 years
  Dietary saturated fat intake, % of total energy intake
Carbohydrate intake | Through study completion, on average 10 years
  Dietary carbohydrate intake, % of total energy intake
Sugar intake | Through study completion, on average 10 years
  Dietary sugar intake, g/day
Fibre intake | Through study completion, on average 10 years
  Dietary fibre intake, g/day
Sodium intake | Through study completion, on average 10 years
  Dietary sodium intake, mg/day
Skipping breakfast | Through study completion, on average 10 years
  Questionnaire measure of regularity of skipping breakfast
Fruit intake | Through study completion, on average 10 years
  Questionnaire measure of regularity of fruit consumption
Vegetable intake | Through study completion, on average 10 years
  Questionnaire measure of regularity of vegetable consumption
Fizzy drink intake | Through study completion, on average 10 years
  Questionnaire measure of regularity of fizzy drink consumption

CONTACTS AND LOCATIONS:
Overall Officials: Seeromanie Harding, PhD, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: Yes
The DASH data are available to researchers via a data request to the MRC Social and Public Health Science Unit. Applications and the data sharing policy for DASH can be found at http://dash.sphsu.mrc.
  ac.uk/DASH_dsp_v1_November-2012_draft.pdf. It reflects the MRC guidance on data sharing with the aim of making the data as widely and freely available as possible while safeguarding the privacy of participants, protecting confidential data, and maintaining the reputation of the study. All potential collaborators work with a link person, an experienced DASH researcher-to support their access to and analysis of the data. The variable-level metadata is available from the study team and also via the MRC Data Gateway.
Supporting Information: Study Protocol, ICF
Time Frame: Data available from 2014 for 10 years.
URL: http://dash.sphsu.mrc.ac.uk

REFERENCES:
- [Result] Harding S, Whitrow M, Maynard MJ, Teyhan A. Cohort profile: The DASH (Determinants of Adolescent Social well-being and Health) Study, an ethnically diverse cohort. Int J Epidemiol. 2007 Jun;36(3):512-7. doi: 10.1093/ije/dym094. Epub 2007 Jul 30. No abstract available. PMID 17664225
- [Result] Lu Y, Sooky L, Silva MJ, Molaodi OR, Karamanos A, Cruickshank JK, Harding S. Longitudinal study of the influence of lung function on vascular health from adolescence to early adulthood in a British multiethnic cohort. J Hypertens. 2017 Nov;35(11):2185-2191. doi: 10.1097/HJH.0000000000001455. PMID 28661960
- [Result] Harding S, Silva MJ, Molaodi OR, Enayat ZE, Cassidy A, Karamanos A, Read UM, Cruickshank JK. Longitudinal study of cardiometabolic risk from early adolescence to early adulthood in an ethnically diverse cohort. BMJ Open. 2016 Dec 14;6(12):e013221. doi: 10.1136/bmjopen-2016-013221. PMID 27979836
- [Result] Faconti L, Silva MJ, Molaodi OR, Enayat ZE, Cassidy A, Karamanos A, Nanino E, Read UM, Dall P, Stansfield B, Harding S, Cruickshank KJ. Can arterial wave augmentation in young adults help account for variability of cardiovascular risk in different British ethnic groups? J Hypertens. 2016 Nov;34(11):2220-6. doi: 10.1097/HJH.0000000000001066. PMID 27490950
- [Result] Harding S, Read UM, Molaodi OR, Cassidy A, Maynard MJ, Lenguerrand E, Astell-Burt T, Teyhan A, Whitrow M, Enayat ZE. The Determinants of young Adult Social well-being and Health (DASH) study: diversity, psychosocial determinants and health. Soc Psychiatry Psychiatr Epidemiol. 2015 Aug;50(8):1173-88. doi: 10.1007/s00127-015-1047-9. Epub 2015 Apr 11. PMID 25861790
- [Result] Whitrow MJ, Harding S. Asthma in Black African, Black Caribbean and South Asian adolescents in the MRC DASH study: a cross sectional analysis. BMC Pediatr. 2010 Mar 25;10:18. doi: 10.1186/1471-2431-10-18. PMID 20334698
- [Result] Harding S, Teyhan A, Maynard MJ, Cruickshank JK. Ethnic differences in overweight and obesity in early adolescence in the MRC DASH study: the role of adolescent and parental lifestyle. Int J Epidemiol. 2008 Feb;37(1):162-72. doi: 10.1093/ije/dym252. Epub 2008 Jan 19. PMID 18204089
- [Result] Maynard MJ, Harding S, Minnis H. Psychological well-being in Black Caribbean, Black African, and White adolescents in the UK Medical Research Council DASH study. Soc Psychiatry Psychiatr Epidemiol. 2007 Sep;42(9):759-69. doi: 10.1007/s00127-007-0227-7. Epub 2007 Jun 29. PMID 17603738
- [Result] Harding S, Maynard MJ, Cruickshank K, Teyhan A. Overweight, obesity and high blood pressure in an ethnically diverse sample of adolescents in Britain: the Medical Research Council DASH study. Int J Obes (Lond). 2008 Jan;32(1):82-90. doi: 10.1038/sj.ijo.0803662. Epub 2007 Jun 19. PMID 17579635
- [Result] Harding S, Maynard M, Cruickshank JK, Gray L. Anthropometry and blood pressure differences in black Caribbean, African, South Asian and white adolescents: the MRC DASH study. J Hypertens. 2006 Aug;24(8):1507-14. doi: 10.1097/01.hjh.0000239285.20315.4d. PMID 16877952